CLINICAL TRIAL: NCT06670105
Title: A Phase 2 Trial of Glofitamab for Minimal Residual Disease in Patients With Large B-cell Lymphoma
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: PI Request
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-1314; NCI-2024-09090 (Other: NCI-CTRP Clinical Trials Registray); NCI-2025-06734 (Other: Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2024-10-31; First posted 2024-11-01 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: B-cell Lymphoma
MeSH Terms: conditions — Lymphoma, B-Cell | interventions — glofitamab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Glofitamab (Experimental): Participants will enter a screening period to determine eligibility for the study
  Interventions: Drug: Glofitamab

INTERVENTIONS:
Drug: Glofitamab — Given by vein

SUMMARY:
The goal of this clinical research study is to learn if glofitamab can help to prevent recurrence of LBCL in patients who have achieved CR after standard first-line therapy but have tested positive for MRD. The safety of glofitamab will also be studied.

DETAILED DESCRIPTION:
Primary Objective:

To determine the rate of undetectable MRD following treatment with glofitamab in patients with LBCL who were MRD positive at the end of standard first line treatment

Secondary Objective:

To determine progression-free survival (PFS), overall survival (OS), and evaluate safety of glofitamab as treatment for patients with LBCL who are MRD positive at end of standard first line treatment

Exploratory Objective:

To determine the biomarkers of response and mechanisms of resistance to glofitamab in LBCL

To determine the kinetics of T-cell activation and exhaustion in patients treated with gofitamab to eliminate MRD

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Histologically diagnosed
* Diffuse large B-cell lymphoma, not otherwise specified (NOS) or
* High grade B-cell lymphoma (NOS or MYC and BCL2 rearrangements) or
* Transformed large B-cell lymphoma from indolent lymphomas (but not Waldenstrom macroglobulinemia/Lymphoplasmacytic lymphoma)
* Have received first line standard of care anthracycline-based chemoimmunotherapy for 6 cycles (with or without 2 more cycles of rituximab) for previously untreated disease
* R-CHOP (cyclophosphamide, doxorubicin, vincristine sulfate, and prednisone)
* DA-EPOCH-R
* Polatuzumab-R-CHP
* Have achieved complete metabolic response by Lugano criteria4 at the end of treatment response evaluation after first line treatment
* MRD Positive at the end of first line treatment
* Performance status ≤2 on the ECOG scale
* Patients must have adequate organ and marrow function as defined below:
* Absolute neutrophil count (ANC) ≥0.5 x 109/L *

  ¡ *Growth factor permitted during screening
* Platelet count ≥50 x 109/L
* Hemoglobin ≥8 g/dL
* Total bilirubin ≤ 3 ULN, unless consistent with Gilbert's
* AST and ALT ≤ 3x upper limit of normal (ULN)
* Alkaline phosphatase < 2.5 ULN
* Creatinine clearance >30 ml/min calculated by modified Cockcroft-Gault formula
* Cardiac ejection fraction ≥ 40%, no evidence of pericardial effusion (except trace or physiological) as determined by an echocardiogram (ECHO), and no clinically significant electrocardiogram (ECG) findings
* All subjects must
* Agree to refrain from donating blood while on study treatment, during dose interruptions and for at least 12 months following the last dose of study treatment.
* Females must agree to abstain from breastfeeding during study participation and for at least 2 months after glofitamab discontinuation.
* The effects of glofitamab on the developing human fetus are unknown. For this reason, women of child-bearing potential and men must agree to use adequate contraception {hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation.

(Refer to Pregnancy Assessment Policy MD Anderson Institutional Policy # CLN1114). This includes all female patients, between the onset of menses (as early as 8 years of age) and 55 years unless the patient presents with an applicable exclusionary factor which may be one of the following:

* Postmenopausal (no menses in greater than or equal to 12 consecutive months).
* History of hysterectomy or bilateral salpingo-oophorectomy.
* Ovarian failure (Follicle Stimulating Hormone and Estradiol in menopausal range, who have received Whole Pelvic Radiation Therapy).
* History of bilateral tubal ligation or another surgical sterilization procedure.
* Females of childbearing potential (FCBP ˜) must:
* Have one negative pregnancy tests via serum or urine prior to starting study therapy. She must agree to ongoing pregnancy testing during the course of the study, prior to day 1 of each cycle, and after end of study therapy. This applies even if the subject practices true abstinence* from heterosexual contact.
* Effective contraception should be used until at least 18 months after pre-treatment with obinutuzumab, 2 months after the last dose of glofitamab, or 3 months after the last dose of tocilizumab (if applicable), whichever is longer.
* Approved methods of birth control are as follows: Hormonal contraception (i.e. birth control pills, injection, implant, transdermal patch, vaginal ring), Intrauterine device {IUD), Tubal Ligation or hysterectomy, SubjecUPartner post vasectomy, Implantable or injectable contraceptives, and condoms plus spermicide. Not engaging in sexual activity for the total duration of the trial and the drug washout period is an acceptable practice; however periodic abstinence, the rhythm method, and the withdrawal method are not acceptable methods of birth control. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.
* Male subjects must:
* Male patients must agree to either remain completely abstinent or use effective contraception from screening until at least 3 months after pre-treatment with obinutuzumab, 2 months after the last dose of glofitamab, 2 months after the last dose of tocilizumab (if applicable), whichever is longer. Men must refrain from donating sperm during this same period.
* Patient must be willing and able to comply with the protocol treatment and procedures.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Having radiologically confirmed relapsed/refractory disease.
* Patients who have not recovered from non-hematological AEs due to prior first line therapy (i.e., have residual toxicities > Grade 1) with the exception of alopecia.
* Known central nervous system lymphoma or leptomeningeal disease.
* Suspicious case at end of treatment from first line treatment should be evaluated with brain MRI with or without lumber puncture.
* Any prior history of other malignancy besides 8-NHL, unless the patient has been free of disease for ≥ 3 years and felt to be at low risk for recurrence by the treating physician, except:
* Adequately treated localized skin cancer without evidence of disease.
* Adequately treated cervical carcinoma in situ without evidence of disease.
* Any life-threatening illness, medical condition, or organ system dysfunction which, in the investigator's opinion, could compromise the subject's safety, or put the study outcomes at undue risk.
* Uncontrolled human immunodeficiency virus (HIV), or active Hepatitis C Virus, or active Hepatitis B Virus infection, or any uncontrolled active significant infection, including suspected or confirmed JC virus infection and SARS-CoV2.
* Patients with inactive hepatitis B infection must adhere to hepatitis B reactivation prophylaxis unless contraindicated. The treatment and monitoring of hepatitis B will follow the institutional standard of practice. Hepatitis B or C serologic status: subjects who are hepatitis B core antibody (anti-HBc) positive and who are surface antigen negative will need to have a negative polymerase chain reaction (PCR). Those who are hepatitis B surface antigen (HbsAg) positive or hepatitis B PCR positive will be excluded. Subjects who are hepatitis C antibody positive will need to have a negative PCR result. Those who are hepatitis C PCR positive will be excluded. Subjects with a history of Hepatitis C who received antiviral treatment are eligible as long as PCR is negative.
* History of severe allergic or anaphylactic reactions or intolerance to anti-CD20 monoclonal antibody therapy or any bispecific antibody.
* History of immunodeficiency (with the exception of hypogammaglobulinemia) or concurrent systemic immunosuppressant therapy (e.g., cyclosporine, tacrolimus, etc., or chronic administration glucocorticoid equivalent of >10mg/day of prednisone) within 28 days of the first dose of study drug with exception of steroid used for IV contrast allergy. In addition, use of inhaled, topical, intranasal corticosteroids or local steroid injection (eg, intra- articular injection) is permitted.
* Clinically significant cardiovascular disease such as uncontrolled or symptomatic arrhythmias, congestive heart failure, or myocardial infarction within 6 months of Screening, or any Class 3 (moderate) or Class 4 (severe) cardiac disease as defined by the New York Heart Association (NYHA) Functional Classification. Subjects with controlled, asymptomatic heart failure during screening can enroll on study.
* History of stroke, seizure disorder or patients requiring antiepileptic therapy or intracranial hemorrhage within 18 months prior to study entry.
* Lactating or pregnant subjects. Pregnant women are excluded from this study for unknown potential for teratogenic or abortifacient effects by glofitamab. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with glofitamab, breastfeeding should be discontinued if the mother is treated with glofitamab. These potential risks may also apply to other agents used in this study.
* Had blood transfusion within 14 days of first dose of study drug.
* Administration of any investigational agent within 28 days of first dose of study drug.
* Patients who have undergone major surgery within 28 days or minor surgery within 3 days of first dose of study drug.
* Administration of a live, attenuated vaccine within 4 weeks before first study treatment administration or anticipation that such a live, attenuated vaccine will be required during the study.
* Patients taking chronic corticosteroids for other diseases, unless administered at a dose equivalent to < 10 mg/day prednisone. For corticosteroids, prednisolone >20 mg daily (or equivalent) qualifies as immunosuppressive and thus is excluded for this use. Note: corticosteroids at any dose are permitted for control of lymphoma-related symptoms, including during screening, and for prophylaxis or AE management during the trial.
* Prior exposure to CD20 x CD3 bispecific antibodies, independently from indication.
* Patients who have concern for the accurate assessment of neuro toxicity.
* Patients who have an active autoimmune disease that has required systemic treatment in past 2 years (i.e., with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered a form of systemic treatment and is allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-06-06 (Estimated); Primary Completion 2030-01-06 (Estimated); Study Completion 2032-01-06 (Estimated)

PRIMARY OUTCOMES:
Safety and Adverse Events (AEs) | Through study completion; an average of 1 year
  Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Dai Chihara, MD,PHD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- The University of Texas M. D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org